CLINICAL TRIAL: NCT01456273
Title: Evaluation of the Efficacy of the Integral Approach (Therapeutic Encounter) Versus the Conventional Medical Approach (Medical Consultation) in Patients With Functional Dyspepsia
Brief Title: From the Biomedical to the Biopsychosocial Model, From Theory to Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Collaborators: Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other)
Responsible Party: Principal Investigator, Fernando Soares Guedes, Professor, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Guedes, FG 01
Record Dates: First submitted 2011-08-23; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Functional Dyspepsia
Keywords: biopsychosocial model; biomedical model; functional dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- A2- Medical consultation + placebo (Placebo Comparator): Traditional medical interview + placebo
  Interventions: Procedure: Traditional Medical Consultation
- B1 - Therapeutic Encounter / Omeprazol (Active Comparator)
  Interventions: Procedure: Therapeutic Encounter
- B2 - Therapeutic Encounter / Placebo (Placebo Comparator)
  Interventions: Procedure: Therapeutic Encounter
- A1- Medical consultation + omeprazole (Active Comparator): Traditional medical interview + omeprazole
  Interventions: Procedure: Traditional Medical Consultation

INTERVENTIONS:
Procedure: Traditional Medical Consultation — Group A will be divided into 2 subgroups : A1- Traditional medical consultation + placebo, and A2- traditional medical consultation plus omeprazole
  Arms: A1- Medical consultation + omeprazole; A2- Medical consultation + placebo
Procedure: Therapeutic Encounter — Group B (who receive care "Therapeutic Encounter") will be divided in subgroup B1, which will receive the "Drug Therapy Classic" and 2 in group B who received placebo.
  Arms: B1 - Therapeutic Encounter / Omeprazol; B2 - Therapeutic Encounter / Placebo

SUMMARY:
This study aims to evaluate, in patients with functional dyspepsia, a model example of medical care based upon the biopsychosocial model (called: the therapeutic encounter) compared with standard medical care based upon the biomedical model (called: medical consultation).

DETAILED DESCRIPTION:
INTRODUCTION Addressing the high costs involved in new medical technology (biotechnology) is a problem that has led individuals and public health services to feel increasingly powerless.

Many authors say that not even an efficient use of resources can ensure better care and health care, a true bottomless pit.

The problem is the conceptual and ideological bases of thinking and acting of the professionals involved. The first misunderstanding is the "narrow approach" and the second is the "process of medicalization."

The curative model and the restricted approach The curative model gets this name because it is not concerned with the causes of the disease process (prevention), only with the effects (the disease). As the effects can be mitigated or even extinct, it is only temporary, because sooner or later they will return with the same format or not, in the same individual or another. It is extremely costly for individuals and for society, because the solutions are palliative. The approach is limited and so are results too.

The process of medicalization Medicalization is the ultimate expression of the distortions of thinking and consequences of the model of health care regulations. It can be understood as the increasingly high dependence on individuals and society overestimating the role that biotechnology could play, and creating a dependency in which one believes that for any problem, regardless of its severity or causal links, there will be a life-saving treatment.

The wrong postures and maintenance of unhealthy habits The model of health care can lead to wrong postures. Many of today's health problems have a direct causal relationship with the passive attitude of individuals, who delegate (to health care and biotechnology) full responsibility for treating their ailments, are reluctant to bring about changes in habits and behaviors because the "curative medicine holds that the doctors can take a magic bullet and get our problems solved."

The strong interest in maintaining the healing model The curative model has a tendency to concentrate on the application of biotechnology to strengthen the multinational pharmaceutical industry and large firms in highly sophisticated biomedical equipment. This has generated a stunning increase of expenditure on health as well as strong interest in this market maintaining its hegemonic space through emphasis on "cure(medicalization of life", rather than the emphasis on prevention and changing habits.

Aim of the study This study will aim to test, in patients with functional dyspepsia, a model example of medical care based upon the biopsychosocial model (called: the therapeutic encounter) compared with standard medical care based upon the biomedical model (called: medical consultation).

What is the biopsychosocial model The biopsychosocial model does not focus exclusively on organic disease. It considers the thinking process of becoming ill with multiple causalities. It tries to understand the man, their psychological, biological, socio-cultural and spiritual interconnections. It argues that the way of being and becoming ill are constructions of the life history of each individual, where the psychological and physiological are inextricably linked. In this perspective, disease becomes an expression of internal conflicts, has a personal character and is linked to the person's relationship with his world (its environment).

This approach has important consequences in medical practice as the doctor's focus of attention shifts to the individual diseases.

The medical care based upon the biopsychosocial model conserves the characteristics of art of medicine. Art in the sense of craftsmanship (the "tailored") as opposed to biomedical technique that is (to systematize, generalize). In fact one must know deeply the technique to apply it with art.

The primary focus continues to be what the patient has in common with others, but in its quirks (it is the art of medicine). It is considered less important if a particular treatment will work, thinking of the majority of patients (the technique), but whether it will work for this particular patient, with his personal problems at the moment of his life in this environment, this location in this country and this region of the world.

Why test it in functional dyspepsia patients

Functional dyspepsia is part of a group of diseases called "Functional Disorders of the Gastrointestinal Tract" that goes beyond the biomedical model:

* They are defined as variable combinations of symptoms, not explained by structural or biochemical changes.
* The diagnostic criteria and parameters for better or worse are based on symptoms reported by patients, this causes some skepticism in the face of more traditional medical view. There are no objective criteria for assessing these disorders.

Why to use placebo

The use of placebo in this study is justified due to the facts:

* Symptoms of functional dyspepsia have a high rate of improvement with placebo. Comparative studies with some drugs show that the placebo effect is up to the order of 30 to 40%.
* can not rule out the placebo effect, if the magnitude of this drug therapies are not compared to placebo.

Justification of the study This study is justified for several reasons, but mainly by the limitations of the biomedical model.

* The changes in the epidemiological profile (which has been occurring in recent decades) are increasingly leaving very clear the role of psychological, socio-cultural and spiritual factors, as expressed by the personality and lifestyle.
* The same biomedicine with its progress and sophistication is showing its inability to provide satisfactory or conclusive answers to many problems, especially for the subjective components that come into greater or lesser degree in any disease.

Biomedicine is too limited in its explanatory power. Many medical professionals realize the psychological reactions of patients and their socioeconomic problems involved in the disease but do not see how to incorporate this information in formulating diagnosis and treatment decisions. The idea of ilness as a phenomenon more or less accidental, originating in the biochemical processes of the body is very restricted, and therefore produces restricted results too.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of functional dyspepsia (according to the Rome II criteria)
* They must be literate so they can read and fill out the questionnaire and a diary of symptoms without the aid of others

Exclusion Criteria:

* Patients who for any reason: not accepting to participate in research, not having signed an informed consent or not answering the questionnaire, the collection period, for whatever reasons
* Abuse or dependence on alcohol, tobacco, medications or other drugs (licit or illicit)
* Diabetes (any type
* pregnancy or breastfeeding (in any stage of the study)
* organic diseases or severe metabolic or evolving (heart disease, severe hypertension, infectious diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Score of dyspeptic symptoms questionnaire administered at the beginning and end of treatment. | between four to six months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fernando S Guedes, Master, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil